CLINICAL TRIAL: NCT01698645
Title: A Spanish , Multicentre, Open-label, Observational Study to Assess Quality of Life and Satisfaction in Subjects Taking PecFent® for the Treatment of Breakthrough Cancer Pain (BTPc)
Brief Title: Patient Satisfaction and Quality of Life Impact - PecFent®
Acronym: Qualipec
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Archimedes Development Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CP070/12
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Breakthrough Cancer Pain
Keywords: quality of life; PecFent; Lazanda; fentanyl; intranasal; breakthrough cancer pain
MeSH Terms: interventions — Fentanyl; Nasal Sprays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PecFent®
  Interventions: Drug: PecFent® (fentanyl) nasal spray

INTERVENTIONS:
Drug: PecFent® (fentanyl) nasal spray

SUMMARY:
National multicenter, prospective, observational study in cancer patients with chronic background pain and breakthrough pain to whom PecFent® has been prescribed under pragmatic condition by a specialist in the treatment of cancer pain conditions.

• Study objectives include assessment of early treatment satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged ≥18 years) with cancer
* Taking at least 60 mg of oral morphine sulfate or equivalent per day for chronic background pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with breakthrough pain
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Satisfaction | Satisfaction will be assessed approximately 1 hour after each breakthrough pain (BTPc) episode treated with PecFent® from completion of titration through Day 7
  Satisfaction will be assessed using a 4-point Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital 12 de Octubre, Madrid, Spain